CLINICAL TRIAL: NCT00139204
Title: An Evaluation of the Effects of Chemotherapy on the Uptake and Retention of Carbon 11 Methionine (C11 MET) in Prostate Cancer, as Assessed by Positron Emission Tomography (PET)
Brief Title: Evaluation of the Effects of Chemotherapy on the Uptake and Retention of Carbon 11 Methionine in Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-419
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Hormone-refractory prostate cancer; PET scan; C11-methionine; positron emission tomography
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Procedure: C11 Methionine PET scan

SUMMARY:
The purpose of this study is to better understand a new type of radiology test called positron emission tomography (PET) with carbon 11 methionine to determine which patients have a beneficial effect from anti-cancer therapy with the drug docetaxel.

DETAILED DESCRIPTION:
In the week before the patients first dose of chemotherapy they will receive a C11 methionine PET scan which takes about 90 minutes. C11 methionine is a radioactively labeled amino acid that is given to the patient intravenously.

Eighteen to twenty days after the patients first dose of docetaxel chemotherapy, they will have another C11 methionine PET scan which is identical to the first scan.

At the end of three cycles of docetaxel chemotherapy (about 2 and 1/2 months on study) another C11 methionine PET scan will be done.

The PET scans will show how well the tumor is taking up methionine.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic hormone-refractory prostate cancer patients who are planned to begin every 3-week docetaxel chemotherapy
* Progression after androgen deprivation therapy
* Serum testosterone < 50ng/ml
* 18 years of age or older

Exclusion Criteria:

* Prior taxane therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-04; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To describe the association between percent change in tumor standardized uptake value (SUV) after c11 methionine administration after one cycle of every three-week docetaxel-based chemotherapy and prostate-specific antigen (PSA) response

SECONDARY OUTCOMES:
To explore the relative value of the change in tumor SUV after C11 methionine administration after one cycle and 3 cycles of docetaxel with respect to PSA progression
to explore optimal cutpoints and measures of SUV change for distinguishing responders from non-responders and progressors from non-progressors and
to evaluate the relationship between the percent change is tumor SUV after C11 methionine administration with freedom from PSA progression in 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts